CLINICAL TRIAL: NCT07178717
Title: A Phase 2, Single-Arm Study of Encorafenib Plus Cetuximab as Rechallenge Treatment of BRAF V600E-mutant Metastatic Colorectal Cancer Patients After Previous Therapy With BRAF Inhibitors-based Combinations: the RefIsh Trial
Brief Title: A Study to Characterize Encorafenib Plus Cetuximab as Rechallenge Treatment for BRAF V600E-mutant Metastatic Colorectal Cancer Patients After Previous Therapy With BRAF Inhibitors-based Combinations
Acronym: REFISH
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Vall d'Hebron Institute of Oncology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VHIO23004; 2023-509564-22-00 (EU CTIS Number)
Record Dates: First submitted 2025-09-02; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Colo-rectal Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — Bevacizumab; encorafenib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Bevacizumab + encorafenib (Experimental)
  Interventions: Drug: Rechalange with bevacizumab + encorafenib

INTERVENTIONS:
Drug: Rechalange with bevacizumab + encorafenib — Patients will receive encorafenib 300mg once daily plus cetuximab 500mg/m2 every 2 weeks until disease progression, unacceptable toxicity, patient request, physician's decision to withdraw treatment, subsequent anticancer therapy or death.

SUMMARY:
This is an open-label, unicentre, single-arm Phase 2 study of encorafenib and cetuximab as rechallenge treatment in patients with BRAF V600E-mutant metastatic colorectal cancer after previous therapy with BRAF inhibitors-based combinations.

The study aims to evaluate the antitumor activity of encorafenib plus cetuximab as a rechallenge strategy measured by progression-free survival rate at 4 months.

Eligible patients (a total of 25) will receive encorafenib 300 mg (four 75 mg capsules) once daily (q.d) in 28-day cycles plus intravenous cetuximab at 500 mg/m2 every 2 weeks (Q2W). Treatment will be administered until progression, unacceptable toxicity, patient request, physician's decision or subsequent anticancer therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of signed and dated informed consent form.
2. Age ≥18 years at the time of informed consent.
3. Histologically- or cytologically confirmed mCRC that is metastatic.
4. Presence of confirmed BRAF V600E mutation.
5. Eligible to receive cetuximab and encorafenib per locally approved label with regard to tumor RAS status.
6. Patients must be previously treated with at least 2 prior regimens for metastatic disease and had demonstrated progressive disease or intolerance to their last regimen. Prior standard chemotherapy must include the following agents: fluoropyrimidine in monotherapy or in combination with irinotecan and/or oxaliplatin with or without anti-VEGF. Combination of chemotherapy with BRAF inhibitor-containing regimen is also permitted.
7. Patients must have received BRAF inhibitor plus anti-EGFR combinations (including but not limited to MEK or ERK inhibitors or chemotherapy) treatment for ≥ 4 months. Patients must have had complete response, partial response or stable disease >6 months during the BRAF inhibitor-based treatment.
8. Patients at study enrollment should have at least 4 months interval since the last administration of BRAF inhibitors.
9. Life expectancy >12 weeks, as determined by the investigator.
10. Patients must have progressed during or within 6 months of the last chemotherapy regimen > Patients who received adjuvant/neoadjuvant chemotherapy and had recurrence during or within 6 months of completion of the adjuvant/neoadjuvant chemotherapy are permitted to count the adjuvant/neoadjuvant therapy as one regimen for advanced disease.
11. Measurable disease according to RECIST v1.1.
12. ECOG performance status 0-1.
13. Adequate bone marrow function characterized by the following at screening:

    1. Absolute neutrophil count (ANC) ≥1.5 x 10^9/L.
    2. Platelets ≥100 x 10^9/L.
    3. Hemoglobin ≥9.0 g/dL (with or without blood transfusions).
14. Adequate hepatic and renal function characterized by the following at screening:

    1. Serum total bilirubin ≤1.5 x upper limit of normal (ULN) and <2 mg/dL. Note: Total bilirubin >1.5 x ULN is allowed if direct (conjugated) ≤1.5 x ULN and indirect (unconjugated) bilirubin is ≤4.25 x ULN.

       Note: Participants with hyperbilirubinemia due to non-hepatic cause (e.g., hemolysis, hematoma) may be enrolled following discussion and agreement with the Sponsor medical monitor.
    2. Alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST) ≤2.5 x ULN, or ≤5 x ULN in the presence of liver metastases.
    3. Adequate renal function defined by an estimated creatinine clearance ≥50 mL/min according to the Cockcroft Gault formula or by 24-hour urine collection for creatinine clearance, or according to local institutional standard method.
    4. Protein < 2+ on dipstick urinalysis or ≤ 1.0 g in a 24-hour urine collection. All patients with ≥2+ protein on dipstick urinalysis at baseline must undergo a 24-hour urine collection for protein.
    5. Adequate electrolytes, defined as serum potassium and magnesium levels within institutional normal limits.

    Note: Replacement treatment to achieve adequate electrolytes will be allowed.
15. Adequate cardiac function characterized by the following at screening:

    • Mean triplicate QT interval corrected for heart rate using Fridericia's formula (QTcF) value ≤480 msec.
16. Able to take oral medications.
17. Highly effective contraception for both male and female subjects if the risk of conception exists during and at least up to 2 months after the last study medication.

Exclusion Criteria:

1. Treatment with another investigational drug or participation in another investigational study at enrolment or within 30 days prior to enrollment.
2. Patient unable to comply with the study protocol owing to psychological, social (lack of social support or social exclusion) or geographical reasons.
3. Patient is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
4. Known history of chronic pancreatitis.
5. Tumors with microsatellite instability or mismatch repair deficiency if they have not received a PD1/PDL1 inhibitor-based treatment, unless medical contraindication.
6. History of chronic inflammatory bowel disease or Crohn's disease requiring medical intervention (immunomodulatory or immunosuppressive medications or surgery) ≤ 12 months before the enrollment in the study.
7. Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following:

   1. History of acute myocardial infarction, acute coronary syndromes (including unstable angina, coronary artery bypass graft [CABG], coronary angioplasty or stenting) ≤ 6 months prior to start of study treatment.
   2. Symptomatic congestive heart failure (i.e., Grade 2 or higher), history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality ≤ 6 months prior to start of study treatment, except atrial fibrillation and paroxysmal supraventricular tachycardia.
8. Impaired hepatic function, defined as Child-Pugh class B or C.
9. Known history of human immunodeficiency virus (HIV), active hepatitis B virus (HBV) infection or active hepatitis C virus (HCV) infection. Patients positive for HCV antibody are eligible only if polymerase chain reaction is negative for HCV RNA. Patients with past exposure to HBV are also eligible for the study provided they are negative for HBV DNA.
10. Has spinal cord compression or clinically active central nervous system metastases, defined as untreated and symptomatic, or requiring therapy with corticosteroids or anticonvulsants to control associated symptoms. Subjects with clinically inactive brain metastases may be included in the study.

    Subjects with treated brain metastases that are no longer symptomatic and who require no treatment with corticosteroids or anticonvulsants may be included in the study if they have recovered from the acute toxic effect of radiotherapy. A minimum of 2 weeks must have elapsed between the end of whole brain radiotherapy and the enrollment in the study.
11. Subjects with leptomeningeal carcinomatosis.
12. Impaired gastrointestinal (GI) function or disease that may significantly alter the absorption of encorafenib (e.g., ulcerative diseases, uncontrolled vomiting, malabsorption syndrome, small bowel resection with decreased intestinal absorption).
13. Knowledge of any other disease or medication that may interfere with study treatment.
14. Presence of any contraindication with regard to the study drugs as specified in the corresponding SmPCs.
15. Patients who achieved progression disease as best response while receiving BRAF inhibitor previously.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-10 (Estimated); Primary Completion 2028-02 (Estimated); Study Completion 2028-08 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | 4 months since the start of treatment
  Progression-free survival rate at 4 months (4-month PFS rate) according to RECIST V1.1 by Investigator assessment.

SECONDARY OUTCOMES:
Progression-free survival | From randomization until the first documented progression, assessed up to 30 months (expected)
  Progression-free survival (PFS) according to RECIST V1.1 by Investigator assessment.
Objective response rate | For the duration of the study, expected 30 months
  Description: Objective Response Rate (ORR) according to RECIST V1.1 by Investigator assessment.
Overal Survival | From date of enrollment until death, up to the duration of the study (expected 30 months)
  Overall survival (OS)
Evaluate the safety and tolerability profile | Through study completion, an average of 1 year
  Incidence and severity of adverse events (AEs), graded by Common Terminology Criteria for Adverse Events (CTCAE) version 5.0. Change in clinical laboratory test parameters, vital signs, ECGs and echocardiogram/MUGA scans.
Clinical efficacy | Through study completion, an average of 1 year"
  Clinical efficacy based on the presence or absence of acquired genomic mechanism of resistance detected in the NGS baseline to the rechallenge.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitari Vall d'Hebron, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No